CLINICAL TRIAL: NCT01077765
Title: Open Label, Multicenter, Single Arm Trial of the Safety and Efficacy of Polyacrylamide Hydrogel Injection in the Management of Human Immunodeficiency Virus-Related Facial Lipoatrophy : THE LIPOPHILL TRIAL
Brief Title: Polyacrylamide Hydrogel Injection in HIV-related Lipoatrophy
Acronym: LIPOPHILL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Mathieu Quintin, Departement clinical research of the developement
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P040601
Record Dates: First submitted 2010-02-26; First posted 2010-03-01 (Estimated); Last update posted 2010-03-01 (Estimated); Status verified 2010-01

CONDITIONS: HIV Infection; Antiretroviral Side Effects; Lipodystrophy Syndrome Related to HIV Infection
Keywords: HIV-associated Lipodystrophy; Polyacrylamide hydrogel
MeSH Terms: conditions — HIV Infections; HIV-Associated Lipodystrophy Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- treatment (Experimental): treatment
  Interventions: Device: Eutrophill

INTERVENTIONS:
Device: Eutrophill — Polyacrylamide Hydrogel

SUMMARY:
Combined antiretroviral therapy (cART) is associated with facial lipoatrophy, which is potentially stigmatizing for HIV-positive patients. Eutrophill is a 2.5% polyacrylamide hydrogel obtained by polymerization of acrylamide monomers with an official half-life of 5 years.

Preliminary encouraging results with the use of polyacrylamide hydrogel for reconstruction of facial lipoatrophy in HIV-infected patients have been previously reported.

The primary objective of the study was to evaluate the long-term efficacy and safety of subcutaneous facial injections of Eutrophill in HIV-infected patients with severe facial lipoatrophy as assessed by facial ultrasonography at screening , after 6, 12 and 24 months

DETAILED DESCRIPTION:
Combined antiretroviral therapy is associated with facial lipoatrophy, which is potentially stigmatizing for HIV-infected patients.

To date, polylactic acid implants (PLA) have been approved for the correction of facial lipoatrophy. The mechanism of action is the increase in new collagen synthesis as a reaction to the presence of the implant in the dermal area. But PLA may be associated with:subcutaneous micronodules and indurations and mid term relapse of lipoatrophy with the need to proceed to new PLA injections EUTROPHILL is a 2.5% polyacrylamide hydrogel with a claimed half-life of 5 years.The gel is relatively viscous and is injected subcutaneously. Following injection, the gel encapsulates. The mechanism of action is the increase in the volume of subcutaneous area by the inert implant

The aim of this multicentric, open-label, single-arm, pilot study was to evaluate the long-term efficacy and safety of intra-dermal facial injections of polyacrylamide hydrogel (EUTROPHILL) in HIV-infected patients with severe facial lipoatrophy. Patients received between 2 and 6 injections every 4 weeks, according to the aesthetic results.

The primary objective of the study was to evaluate the long-term efficacy of subcutaneous facial injections of EUTROPHILL in HIV-infected patients with severe facial lipoatrophy as assessed by facial ultrasonography at screening , after 6, 12 and 24 months

The secondary objectives of the study were:

to evaluate the clinical efficacy by facial photography at screening, after 6, 12 and 24 months; to evaluate Overall Treatment Satisfaction according to patients , close relatives and physicians ; to evaluate changes in quality of life (ABCD questionnaire) ABCD questionnaire is a specific questionnaire validated for HIV-infected patients suffering from lipodystrophy; to evaluate changes in patient's anxiety and depression (HADS questionnaire); to evaluate the safety of the infiltration techniques;

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected patients
* 18 years of age or older
* Severe facial lipoatrophy.
* Stable antiretroviral treatment at least 3 months prior to the inclusion
* CD4 cell count > 100 cells/mm3
* Written informed consent

Exclusion Criteria:

* History of surgical or cosmetic intervention for facial lipoatrophy
* Ongoing opportunistic infection
* Any facial skin disease including Kaposi Sarcoma
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-11; Primary Completion 2008-07 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Cutaneous tissue thickness of the cheeks assessed by facial ultrasonography | 12 months

SECONDARY OUTCOMES:
Facial photography at screening,Overall Treatment Satisfaction according to patients close relatives and physicians,Changes in quality of life (ABCD questionnaire) after Changes. | 6, 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Piketty, Principal Investigator — Assistance Publique Hôpitaux de Paris-HEGP
Locations (1):
- Hopital europeen Georges Pompidou, Paris, France